CLINICAL TRIAL: NCT01527734
Title: COMPARISON OF THE PHARMACOKINETICS AND SAFETY OF LIQUID (30 µg) AND LYOPHILIZED TETRODOTOXIN (15 µg AND 30 µg) FOLLOWING SINGLE AND TWICE DAILY SUBCUTANEOUS DOSE ADMINISTRATION TO HEALTHY VOLUNTEERS-DETERMINATIONS IN BLOOD AND URINE
Brief Title: Comparison Study of Liquid and Lyophilized Formulations of Subcutaneous Tetrodotoxin (TTX) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wex Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Screening
Other Study IDs: TTX-CINP-201PK
Record Dates: First submitted 2012-01-23; First posted 2012-02-07 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: Comparison study
MeSH Terms: interventions — Tetrodotoxin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo
- Tetrodotoxin, TTX (Experimental)
  Interventions: Drug: Tetrodotoxin

INTERVENTIONS:
Drug: Tetrodotoxin — 15ug and 30ug once or twice a day for 1 or 2 days.
  Arms: Tetrodotoxin, TTX
Drug: placebo — 1ml once or twice a day for 1 or 2 days.
  Arms: Placebo

SUMMARY:
The study design is a randomized, double-blind, placebo-controlled, parallel-group, dose comparison with a open-label, crossover, formulation comparison.

ELIGIBILITY:
Inclusion Criteria:

* Normal renal function

Exclusion Criteria:

* History of multiple clinically significant drug allergies

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2011-12; Primary Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Compare plasma and urine PK profiles of TTX following doses of Lyophilized and Injectable Liquid TTX | 26 timepoints over 48 hours
  PK timepoints occurred at 0,0.33,0.67,1, 1.5,2,4,6,8,10,12,14 and 24 hours after first dose on Days 1 & 2. Liquid and Lyophilized formulations will be assessed using ANOVA of the T-R ratio based on log-transformed AUC and Cmax values.

SECONDARY OUTCOMES:
Assess the safety and tolerability of TTX following the administration of Lyophilized and Liquid TTX | signage of the ICF to Day 10
  Safety was assessed through the collection of AE's, concomitant medications, clinical laboratory assessments, neurological assessments and vital signs. Where summary statistics are presented, these will include n, mean, standard deviation, median, minimum, and maximum.

CONTACTS AND LOCATIONS:
Locations (1):
- Comprehensive Clinical Research, Tacoma, Washington, United States

REFERENCES:
- See also: Sponsor website — http://www.wextech.ca/